CLINICAL TRIAL: NCT07032324
Title: A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell Therapy, in Patients With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Clinical Study Exploring CT1190B in the Treatment of Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma ( CT1190B-CG1101 )
Acronym: CT1190B
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qian Wenbin (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Qian Wenbin, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1190B-CG1101_01
Record Dates: First submitted 2025-06-09; First posted 2025-06-23 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
Keywords: CT1190B
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: B-Cell Non-Hodgkin Lymphoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): CT1190B and CT1190B-P cells infusion
  Interventions: Drug: CAR T cells

INTERVENTIONS:
Drug: CAR T cells — chimeric antigen receptor T cells

SUMMARY:
A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell therapy, in Patients with Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose exploratory clinical study to evaluate the safety, efficacy, cellular pharmacokinetics, and pharmacodynamics of CT1190B cells in patients with B-NHL. It is planned to enroll 6-24 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the study visit schedule and other protocol requirements and agree to be in long term follow-up (LTFU) for up to 15 years as mandated by the regulatory guidelines.
2. 18-75 years old;
3. Histologically or cytologically confirmed B-NHL, according the 5th edition of the WHO classification of haematolymphoid tumours, including:

1) Cohort A1: Large B-cell lymphoma, including diffuse large B-cell lymphoma not other specified (DLBCL, NOS), primary mediastinal large B-cell lymphoma (PMBCL), high-grade B-cell lymphoma, transformed follicular large B-cell lymphoma (FLBL)/Grade 3b follicular lymphoma ( FL) 2) Cohort A2: Mantle cell lymphoma (MCL); 3) Cohort B1: Grade 1 ~ 3a FL; 4) Cohort B2: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) according to iwCLL2018 diagnose criteria , with the exception of participants who are currently transformed into Richter 's syndrome; 4. Previous treatment requirement: 5) Cohort A1: Previously received at least 2 lines of systemic therapy, including anti-CD20 drugs (unless the investigator had determined that the tumor is/is CD20 negative) and anthracycline containing regimens, anti-CD20 drugs maintenance alone will not be counted as 1 line of treatment; for participants with transformed FL (FLBL), any treatment administered prior to transformation will not be counted as a prior line.

6) Cohort A2: at least 2 prior lines of systemic therapy, including anthracycline- or bendamustine-containing chemotherapy, anti-CD20 drugs ( unless the investigator had determined that the tumor is/is CD20 negative) and a BTK inhibitor; and CD20 monoclonal antibody alone will not be count as 1 line of treatment; 7) Cohort B1: previously received at least 2 lines of systemic therapy, including anti-CD20 drugs ( unless the investigator had determined that the tumor is/is CD20 negative) and anthracycline-containing chemotherapy regimens, and CD20 monoclonal antibody alone will not be counted as 1 line of treatment; 8) Cohort B2: at least 2 prior lines of therapy, including immunotherapy or chemotherapy and a BTK inhibitor, or BTK inhibitor who are not suitable for immunotherapy or chemotherapy

5. Intolerance to last treatment, or have progressed on or after the last treatment and currently require therapy.

6. At least one of the following:

1) CT testing: Intranodal lesions > 1.5 cm in long diameter, or Extranodal lesions > 1.0 cm in long diameter, 2) PETCT testing: [18F] fluorodeoxyglucose (FDG) positron emission tomography (PET) positive lesion per Lugano criteria at screening (Deauville score 4 or 5) 3) CLL participants requiring treatment according to iwCLL criteria (refer to Appendix 4); 7. Expected survival > 12 weeks; 8. Eastern Cooperative Oncology Group (ECOG) score 0-1; 9. Participants should meet the following test results

1. CBC: ① platelet (PLT) ≥ 75 × 10 9/L (for participants with bone marrow or peripheral blood involvement: PLT ≥ 50 × 10 9/L), ②hemoglobin (Hb) ≥ 80 g/L (for participants with bone marrow or peripheral blood involvement: Hb ≥ 60 g/L);
2. Endogenous creatinine clearance ≥ 30 mL/min (using the Cockcroft -Gault formula);
3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN and total bilirubin ≤ 1.5 × ULN ; if there is liver involvement: AST and ALT ≤ 5 × ULN and total bilirubin ≤ 3.0 × ULN ;
4. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

10. Female participants of childbearing potential must have a negative pregnancy test at screening and prior to receiving preconditioning therapy and are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating eggs for 1 year after receiving study treatment infusion during the study; male participants are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment if they are sexually active with a female of childbearing potential. Sperm donation is absolutely prohibited for 1 year after receiving study treatment infusions during the study for all male participants.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Has HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (HCV antibody and HCV-DNA positive);
3. Has any current uncontrolled active infection, including but not limited to participants with active tuberculosis (investigator 's judgment);
4. Participants' toxicities caused by previous treatment did not recover to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator;
5. Autologous stem cell transplantation within 12 weeks prior to signing informed consent;
6. Prior therapy targeting CD19 (unless CD19 or CD20 target remains positive) ;
7. Has received treatment for the disease within 14 days before FC, including but not limited to cytotoxic therapy, monoclonal antibodies or ADCs, targeted therapy, radiotherapy, epigenetic therapy, or investigational agents, or invasive investigational medical devices within 14 days before informed consent. If the radiation field covers ≤ 5% of the bone marrow reserve, the participant is eligible regardless of the end date of radiotherapy;
8. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids;
9. Vaccination with live attenuated vaccines, inactivate vaccines or RNA vaccines within 4 weeks prior to informed consent;
10. Participants who are allergic or intolerant to preconditioning drugs, tocilizumab, or allergic to the components (DMSO) in CT1190B cell infusion preparation; or have other previous history of severe allergy such as anaphylactic shock;
11. Participants with any of the following cardiac conditions within 6 months prior to screening:

1) New York Heart Association (NYHA) Class III or IV heart failure; 2) Myocardial infarction, coronary artery bypass graft surgery, or unstable angina within 6 months before screening; 3) History of clinically significant uncontrolled arrhythmia, e.g., ventricular arrhythmia; 4) History of severe non-ischemic cardiomyopathy; 5) Left ventricular ejection fraction (LVEF) < 45% as assessed by echocardiogram or multimodal acquisition (MUGA) scan; 6) Other cardiac diseases that, in the opinion of the investigator, may jeopardize the participant 's well-being due to participation in this clinical study; 12. Oxygen saturation < 92%, or suffering from other serious lung diseases, which may endanger the participant 's life as judged by the investigator; 13. Presence of a second primary malignancy requiring treatment or not in complete remission within the past 2 years, except for the following successfully treated tumors with low malignancy such as non-metastatic basal cell or squamous cell skin cancer, non-metastatic prostate cancer, breast or cervical carcinoma in situ, non-muscle-invasive bladder cancer, or thyroid cancer; 14. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract); 15. Participants are unable or unwilling to comply with the requirements of the study protocol or are otherwise unsuitable for participating in this clinical study in the investigator 's assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07-08 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT1190B/CT1190B-P infusion | 12 months after CT1190B/CT1190B-P infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria.
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT1190b/CT1190b-p infusion

SECONDARY OUTCOMES:
Overall response rate#ORR# | Evaluate at 4, 8, 12 weeks and 6,9,12month after CAR-T infusion]
  The proportion of patients with complete remission #CR# /partial response (PR) after CT1190B/CT1190B-P infusion.
Complete response rate (CRR) | 12 months after CT1190B/CT1190B-P infusion
  The proportion of patients with complete response(CR) after CT1190B/CT1190B-P infusion
Duration of remission(DOR) | 12 months after CT1190B infusion
  Participants achieving CR/PR will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Progression-free survival (PFS) | 12 months after CT1190B infusion
  The time from the infusion of CT1190B cells to the first assessment of disease progression or death.
Overall survival (OS) | 12 months after CT1190B infusion.
  defined as the time from the date of receiving the infusion to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: qian wenbin MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No